CLINICAL TRIAL: NCT04165525
Title: ConMed HelixAR™ ElectroSurgical Generator With Argon Beam Coagulation Technology (CHEST) Study
Brief Title: ConMed HelixAR™ ElectroSurgical Generator With Argon Beam Coagulation Technology Study
Acronym: CHEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SurgiQuest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DD01112019
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-05

CONDITIONS: Mastectomy; Lymphedema
Keywords: comparison of ablation devices
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Intervention Model Description: Perspective, randomized, concurrently controlled
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HelixAR Electrosurgical Generator (HEG) (Active Comparator): Argon gas and high frequency electrical current ablation device
  Interventions: Device: Ablation
- Conventional Electrosurgical Coagulation (CEC) Systems (Active Comparator): Standard Bovie electrosugical device without argon gas
  Interventions: Device: Ablation

INTERVENTIONS:
Device: Ablation — comparison of using an argon gas and high frequency electrical current ablation device with a standard Bovie electrosugical device without argon gas.

SUMMARY:
A PROSPECTIVE, RANDOMIZED, CONTROLLED STUDY TO EVALUATE DEVICE EFFICACY BETWEEN THE HELIXAR ELECTROSURGICAL GENERATOR (HEG) VS. CONVENTIONAL ELECTROSURGICAL COAGULATION (CEC) FOR CUTTING AND/OR COAGULATION OF TISSUE DURING MASTECTOMY PROCEDURES

DETAILED DESCRIPTION:
The objective of this study is to evaluate device efficacy between the HelixAR Electrosurgical Generator (HEG) and Conventional Electrosurgical Coagulation (CEC) Systems for cutting and/or coagulation of tissue during mastectomy procedures and reconstructive surgery.

The study is designed and powered to demonstrate the superiority of the HEG to CEC in relation to a key efficacy measure: post-mastectomy procedure time to hemostasis. Secondary outcome measures include: infection, drain duration, total drain output, blood loss, and device related adverse events. These outcomes will be evaluated in a controlled population undergoing mastectomy procedures.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 80 years of age;
2. Capable and willing to give informed consent;
3. Acceptable candidate for a unilateral or bilateral mastectomy and reconstruction. All subjects enrolled and consented will undergo mastectomy with a breast reconstruction procedure, if it is in the subject's best interest.

Exclusion Criteria:

1. Advanced refusal of blood transfusion, if necessary;
2. Active systemic or cutaneous infection or inflammation;
3. Pre-existing immunodeficiency disorder and/or chronic use of systemic steroids;
4. Uncontrolled diabetes mellitus
5. Known, significant history of bleeding diathesis, or coagulopathy, or Von Willebrand's disease or current platelet count < 100,000 cells/mm3, or baseline INR ≥1.8, or fibrinogen level less than 150 mg/dl (if received a fibrinolytic agent within prior 24 hours);
6. Severe co-existing morbidities having a life expectancy of less than 30 days;
7. Currently involved in any other investigational clinical studies that could influence outcomes;
8. Significant anemia with a hemoglobin level less than 10 g/dL or a hematocrit less than 30%;
9. Renal insufficiency (serum creatinine of > 2.5 mg/dl);
10. Females who are pregnant, planning to become pregnant within 3 months of the procedure, or lactating;
11. Patients who have had previous partial mastectomies with scar tissue affecting the area to be resected.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
The time measured from post-mastectomy to hemostasis for each operated breast. | Inter-operative
  time

SECONDARY OUTCOMES:
drain output | up to two weeks post surgery
  ml

OTHER OUTCOMES:
infection rate | two months from procedure
  comparison between arms

CONTACTS AND LOCATIONS:
Overall Officials: Stacey A Carter, MD, Principal Investigator — Baylor St. Luke's Medical Center
Locations (1):
- Baylor St. Luke's Medical Center, Houston, Texas, United States

REFERENCES:
- [Background] McGuire A, Brown JA, Malone C, McLaughlin R, Kerin MJ. Effects of age on the detection and management of breast cancer. Cancers (Basel). 2015 May 22;7(2):908-29. doi: 10.3390/cancers7020815. PMID 26010605
- [Background] Steiner, C.A.; Weiss, A.J.; Barrett, M.L.; Fingar, K.R.; Davis, P.H (2016).
- See also: Breast cancer statstical facts — https://seer.cancer.gov/statfacts/html/breast.html